CLINICAL TRIAL: NCT00095485
Title: Impact of Move to CRC on Physical Activity of Employees
Brief Title: Impact of Move to Clinical Research Center on Physical Activity of Employees
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 050027; 05-CC-0027
Record Dates: First submitted 2004-11-05; First posted 2004-11-08 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-11

CONDITIONS: Healthy
Keywords: Activity Level; Musculoskeletal; Healthy Volunteer; Physical Activity
MeSH Terms: conditions — Motor Activity

SUMMARY:
This study will examine the changes that the move from NIH's Building 10 Clinical Center (CC) into the Clinical Research Center (CRC) may have on the amount of activity a person engages in daily, as registered by a pedometer, which measures horizontal and vertical steps. The investigators in this study hope to better understand the impact that the move will have had on one group of employees compared with the impact for other groups. Moving to a new work location may require physical activity that is different from what employees currently experience on the job. In the new location, they may be walking longer or shorter distances; they may also be climbing fewer or more stairs. In addition, they may need to walk more quickly to accomplish the same tasks. It is important to understand how the move from the CC to the CRC influences employees' health, well-being, and overall function. Physical measures, such as blood pressure, will be examined. So will how well employees are adjusting to the new location-for example, through information about work-related injuries.

Clinical Center employees who are able to walk, whose move dates allow 10 days in the Clinical Center before the move, who wish to participate in the study and are able to wear a pedometer, and whose work requirements include a sufficient amount of walking may be eligible for the study.

Participants will undergo the following procedures before the move into the CRC and then 1 month after the move. Each evaluation will take about 30 minutes:

* Brief history about age, medical problems, and current medications.
* Measurements of heart rate, blood pressure, height, and weight.
* Completing a brief questionnaire about the history of injuries, such as back pain, tendonitis, and bursitis.

In addition, participants will complete a questionnaire about daily life and leisure activities, consisting of 94 questions, to take about 20 minutes to complete. There will also be a measurement of the distance that participants can walk in 2 minutes.

A pedometer will be provided to each participant and will remain the property of that person. Participants will receive a daily log on which to record the number of steps they have walked and the distance as registered by the pedometer. About 5 minutes a day will be needed to record such information. The information that participants provide will be coded. They will not be personally identified, nor will the information be discussed with other people, including supervisors or co-workers.

Information collected will be analyzed for changes in activity patterns and will be analyzed by groups of staff. For example, the investigators may wish to compare the activity of nurses before and after the move and then compare that information with information collected from food service workers, or personnel serving as messengers or escorts. Participants may find the information gathered to be useful to them as individuals. That is, they may learn that their activity has increased as a result of the move to the new location. They may have benefited by having lost weight or lowered their blood pressure.

DETAILED DESCRIPTION:
This project attempts to answer three questions about employees in the Magnuson Clinical Center. It is designed to study the effects of the move into the CRC on the amount of activity an individual performs daily in terms of units measured by a waist mounted pedometer (horizontal and vertical steps).

The hypotheses are:

1. There will be an increase in amount of activity in CRC compared with CC (horizontal distance traveled, up/down activity including stairs and chairs).
2. There will be an increase in walk velocity after move into CRC. This implies an increased level of aerobic capacity.

There will be an increase in the musculoskeletal symptoms, especially in the lower extremities and low back after move to the CRC. This implies there will be overuse of lower extremities because of increased activity.

ELIGIBILITY:
Inclusion Criteria:

Any CC employee who is ambulatory, whose move date allows 10 days in CC prior to move, who wishes to participate in the study and whose work requirements include sufficient amount of walking so that they are not primarily confined to one office module.

Exclusion Criteria:

1. inability to wear a pedometer; and record pedometer data
2. musculoskeletal impairments that significantly limit ambulation, e.g. recent fractures, tendinitis

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150
Dates: Start 2004-11; Study Completion 2005-11

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center (CC), Bethesda, Maryland, United States